CLINICAL TRIAL: NCT06673589
Title: Brain-to-brain Synchrony as a Mechanism of Field Effects of Consciousness
Brief Title: Brain-to-brain Synchrony in Ss With Different Levels of Social Interaction
Status: Recruiting | Type: Observational
Sponsor: Maharishi International University (Other)
Responsible Party: Principal Investigator, Fred Travis, Professor, Director of the Center for Brain, Consciousness and Cognition, Maharishi International University
Other Study IDs: MIU 001
Record Dates: First submitted 2024-06-17; First posted 2024-11-05 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Social Dynamics
Keywords: Consciousness; Hyper-scanning; Social Neuroscience
MeSH Terms: interventions — Meditation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Social Entanglement: Couples, good friends and strangeers
  Interventions: Behavioral: Transcendental Meditation
- good friends from the same region of the country: Plus, extensive social interaction--daily
  Interventions: Behavioral: Transcendental Meditation
- strangers from different countries: Interact minimally--less than once/week
  Interventions: Behavioral: Transcendental Meditation

INTERVENTIONS:
Behavioral: Transcendental Meditation — meditation practice

SUMMARY:
Brain-to-brain synchrony will be measured between pairs of subjects with different levels of similarity of DNA and social interactions

DETAILED DESCRIPTION:
Brain-to-brain synchrony will be measured in five pairs of identical twins, five pairs who are good friends and from the same region of a country, and five pairs of strangers from different countries when they practice Transcendental Meditation practice

ELIGIBILITY:
Inclusion Criteria:

* healthy fit the cohort criteria practice TM

Exclusion Criteria:

* mental or physical issue

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy adult population that practices TM
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Brain-to-Brain Synchrony | 20 minute TM
  EEG (electroencephalography) coherence between 32 sensors in the 10-10 System in all frequency bands

SECONDARY OUTCOMES:
Tracing of depth of meditation (This is a graphic measure.) | after 20 minute meditation
  Use a line to indicate depth of meditation

CONTACTS AND LOCATIONS:
Overall Officials: Fred Travis, PhD, Principal Investigator — Maharishi International Uniersity
Locations (1):
- Maharishi International University, Fairfield, Iowa, United States

IPD SHARING:
Plan to Share IPD: Undecided
We are planning how to store 200 MB files in BDF format on a server